CLINICAL TRIAL: NCT04194463
Title: Maintaining Fitness During Neo-adjuvant Chemotherapy for Oesophago-gastric Cancer: a Feasibility Study to Design and Investigate the Utility of a Simple, Home-Based, Exercise Intervention During Chemotherapy. (ChemoFit)
Brief Title: Maintaining Fitness During Neo-adjuvant Chemotherapy for Oesophago-gastric Cancer: a Feasibility Study
Acronym: ChemoFit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09041
Record Dates: First submitted 2019-10-01; First posted 2019-12-11 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Adenocarcinoma; Gastric Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ChemoFit exercise prehabilitation intervention (Experimental): Exercise intervention consisting of walking and increasing daily step count. This is monitored by wearing a pedometer device. Other part of intervention are 5 simple strengthening exercises.
  Interventions: Other: ChemoFit exercise prehabilitation intervention

INTERVENTIONS:
Other: ChemoFit exercise prehabilitation intervention — Exercise intervention consists of walking monitored by wearing a pedometer device. After a baseline measurement of participant's walking activity is done, increase in step count from baseline step count is prescribed. This increase in step count is achieved by walking or jogging at moderate intensity for a target of 30 minutes per day, each day. Participants are also encouraged to perform other physical if they wish and are able to. Patients are regularly contacted by a member of the research team on a weekly basis and given an option to maintain or to increase their step count further. The same approach is used after each week of the intervention. Strengthening exercises will form a further part of the exercise intervention. They are performed every day, 7 days a week. Patients are supplied with resistance bands with handles. They are educated on how to perform two repetitions of 5 simple exercises, each for 1 minute duration.

SUMMARY:
Feasibility study to investigate the utility of a simple, home-based, exercise intervention during and after neo-adjuvant chemotherapy but prior to surgery for esophageal and gastric adenocarcinoma.

DETAILED DESCRIPTION:
The principle aim of this study is to test the feasibility of utilising a home-based 'prehabilitation' exercise regimen in oesophago-gastric patients during preoperative chemotherapy and the period leading up to surgical resection. The investigators also hope to explore secondary outcomes of such a regimen, such as maintenance of fitness, the incidence of sarcopenia, muscle function and the outcomes of therapy. The investigators will explore the added value of blood-borne frailty biomarkers to objectively measure changes in physiology during neo-adjuvant chemotherapy (NAC). This will be tested using CPET, CT measured sarcopenia, grip strength and a small panel of biomarkers as secondary outcome and exploratory measures. Thus the main question is: 'Will patients participate in a home-based exercise programme during and after NAC for oesophago-gastric cancer?'

ELIGIBILITY:
Inclusion Criteria:

* Operable adenocarcinoma of the oesophagus, oesophago-gastric junction and stomach (locally advanced adenocarcinoma with planned preoperative chemotherapy, T3+, T1/2 N+)
* Planned preoperative chemotherapy with ECX, ECX variant or FLOT chemotherapy
* Age >18
* Ability to complete CPET
* Ability to consent to study and carry out the planned intervention.

Exclusion Criteria:

* Standard contraindications to CPET testing as defined by ATS Guidance
* Orthopaedic limitations to CPET and / or daily exercise, for example, amputation, severe knee or hip disease.
* Inoperable cancer at initial screening MDT
* Planned non-surgical treatment with either radiotherapy or combined chemoradiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Defined as the proportion of all patients approached that agree to enter the study.
Completion rate | 1 year
  Defined as the proportion of all patients that enter the study that remain participants at the end of the defined study period (at surgery).
Individual compliance | 1 year
  With the intervention, defined as the percentage of intervention days when the patient was wearing his/her pedometer, was contactable every week and was recording his/her daily step count.

SECONDARY OUTCOMES:
CPET measurements | 1 year
  Cardiopulmonary fitness measured by cardiopulmonary exercise testing.
Sarcopenia | 1 year
  Change in amount of L3 level skeletal muscle area
Sarcopenia | 1 year
  Change in grip strength
Step count | 1 year
  Change in daily step count from pedometer each day
Quality of life | 1 year
  Quality of life using QLQ-C30 and QLQ-OG25 questionnaires
End of study questionnaire | 1 year
  Subjective perception of intervention using questionnaire
Focus group | 1 year
  End of study 'PPI' focus group to assess exercise intervention
Outcome of oncology treatment | 1 year
  Percentage of planned chemotherapy delivered
Outcome of oncology treatment | 1 year
  Number of patients with dose reductions or who terminate chemotherapy early
Outcome of oncology treatment | 1 year
  Admissions to hospital with chemotherapy induced toxicity

OTHER OUTCOMES:
Exploratory outcome measures | 1 year
  Circulating biomarkers that measure frailty and immune function

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Infirmary, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Cooper M, Chmelo J, Sinclair RCF, Charman S, Hallsworth K, Welford J, Phillips AW, Greystoke A, Avery L. Exploring factors influencing uptake and adherence to a home-based prehabilitation physical activity and exercise intervention for patients undergoing chemotherapy before major surgery (ChemoFit): a qualitative study. BMJ Open. 2022 Sep 22;12(9):e062526. doi: 10.1136/bmjopen-2022-062526. PMID 36137639
- [Derived] Chmelo J, Phillips AW, Greystoke A, Charman SJ, Avery L, Hallsworth K, Welford J, Cooper M, Sinclair RCF. A feasibility trial of prehabilitation before oesophagogastric cancer surgery using a multi-component home-based exercise programme: the ChemoFit study. Pilot Feasibility Stud. 2022 Aug 9;8(1):173. doi: 10.1186/s40814-022-01137-6. PMID 35945625
- [Derived] Chmelo J, Phillips AW, Greystoke A, Charman SJ, Avery L, Hallsworth K, Welford J, Sinclair RCF. A feasibility study to investigate the utility of a home-based exercise intervention during and after neo-adjuvant chemotherapy for oesophago-gastric cancer-the ChemoFit study protocol. Pilot Feasibility Stud. 2020 Apr 23;6:50. doi: 10.1186/s40814-020-00597-y. eCollection 2020. PMID 32346484